CLINICAL TRIAL: NCT04607993
Title: Study on the Effectiveness and Feasibility of Prone Position Ventilation Technique for Postoperative Acute Lung Injury in Infants With Congenital Heart Disease
Brief Title: Study on the Effectiveness and Feasibility of Prone Position Ventilation Technology in Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNF202043
Record Dates: First submitted 2020-10-28; First posted 2020-10-29 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-02

CONDITIONS: Investigative Techniques

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone position ventilation technique (Experimental): Prone position ventilation for children with congenital heart disease after surgery
  Interventions: Behavioral: Prone position ventilation technique
- Control group (No Intervention): conventional postoperative position, no prone position ventilation

INTERVENTIONS:
Behavioral: Prone position ventilation technique — 1. Inform the children's family members of the purpose and method of prone position ventilation
  2. Assess the fixation of various catheters
  3. Suspend feeding before placing prone position
  4. Confirm the time to start prone position ventilation under the joint assessment of medical staff
  5. Place the child in a prone position with the participation of researchers, doctors and nursing staff, with the child's head tilted to one side to avoid damage to the eyes and nose due to compression, and the arms are bent upward to form a "W" . Bend both lower limbs downward to form an "M" shape, and use a soft pillow cushion to measure the knee joints to avoid compression
  6. The whole process ensures the smooth fixation of tracheal intubation and various catheters
  7. Proper sedation during prone position ventilation to achieve good human-machine synchronization
  8. At least 6-8 hours in prone position every day
  Arms: Prone position ventilation technique

SUMMARY:
The purpose of this study was to compare the effects of conventional lying position and prone position ventilation on infants with acute lung injury after surgery for congenital heart disease. To explore the effectiveness and feasibility of prone position ventilation for children with acute lung injury after congenital heart disease surgery.

DETAILED DESCRIPTION:
The prone position has been used to treat severe hypoxemia in patients with acute respiration dysfunction syndrome (ARDS) since the 1970s, and it has significant effectiveness in improving gas exchange. Acute lung injury (ALI) is a common complication after congenital heart disease. The clinical manifestation is refractory hypoxemia. At present, mechanical ventilation is one of the main methods for the treatment of acute lung injury-induced respiratory distress syndrome. Prone position ventilation refers to placing the patient in the prone position during mechanical ventilation to expand the lungs in the atelectasis area and improve the ratio of lung ventilation and perfusion.

Prone position ventilation technology as an important lung protection ventilation strategy has been widely used clinically at home and abroad. Compared with adults, children are more convenient and easy to implement. Due to the exact mechanism of improving oxygenation function, the current domestic and foreign development of pediatric prone ventilation technology is mainly focused on children with ARDS. There are few studies on high-quality application effects after pediatric cardiac surgery, and almost no research has been carried out, especially for pediatric heart The indications for the implementation of the prone position after the disease surgery, the specific standardized process including the position angle, the prone duration plan, etc. all need to be studied. Therefore, there is an urgent need to develop prone position ventilation technology for critically ill children with congenital heart disease after surgery to reduce postoperative pulmonary complications and shorten the time of mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lung injury after congenital heart disease or chest X-ray CT suggest that pulmonary complications need to strengthen body drainage
* Establish artificial airway, such as tracheal intubation
* Children aged 0-12 months
* Stable hemodynamics, more than 72 hours after surgery
* Informed consent of family members

Exclusion Criteria:

* Unstable hemodynamics, severe hypotension, ventricular arrhythmia
* Intracranial hypertension
* Active acute bleeding
* Spinal injuries and untreated unstable fractures, orthopedic surgery or recent abdominal surgery
* Facial trauma
* Severe pneumothorax
* Delayed chest closure and wound infection, children who need to be immobilized

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Oxygenation index | at 6th hours after enrollment
  Oxygenation index refers to a goal in respiratory therapy,OI(mmHg)=PaO2/FiO2 It is a continuous variable.

SECONDARY OUTCOMES:
Lung compliance | at 6th hours after enrollment
  Lung compliance refers to the change in lung volume caused by a change in unit pressure, which represents the impact of changes in chest pressure on lung volume. It would be obtained by ventilator . It is a continuous variable. Its unit is ml/cmH2O.

CONTACTS AND LOCATIONS:
Overall Officials: xu yulu, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- CICU, Cardiovascular Center, Childrens Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu YL, Mi YP, Zhu MX, Ren YH, Gong WJ, Fu WJ, Wang HM, Ye L, Wang Y, Zhou XY, Chen Y, Chen YY, Gu LQ, Gu Y, Jia B, Hu J, Hu XJ. Feasibility and effectiveness of prone position ventilation technique for postoperative acute lung injury in infants with congenital heart disease: study protocol for a prospective randomized study. Trials. 2021 Dec 18;22(1):929. doi: 10.1186/s13063-021-05895-1. PMID 34922610